CLINICAL TRIAL: NCT04944069
Title: Almonertinib Combined With Bevacizumab for EGFR-Mutant NSCLC Patients With Leptomeningeal Metastasis: A Prospective, Open-label, Multi-center, Single-arm Study
Brief Title: Almonertinib With Bevacizumab for EGFR-Mutant NSCLC Patients With Leptomeningeal Metastasis
Acronym: ATTRACT
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HSM-10296-A016
Record Dates: First submitted 2021-05-26; First posted 2021-06-29 (Actual); Last update posted 2021-06-29 (Actual); Status verified 2021-05

CONDITIONS: NSCLC; Leptomeningeal Metastasis; EGFR Activating Mutation
Keywords: Leptomeningeal Metastasis; Non-Small Cell Lung Cancer; EGFR Activating Mutation; Almonertinib; Bevacizumab
MeSH Terms: conditions — Meningeal Carcinomatosis; Carcinoma, Non-Small-Cell Lung | interventions — aumolertinib; Bevacizumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Almonertinib With Bevacizumab (Experimental): Almonertinib 110 mg oral once daily with Bevacizumab 15 mg/kg intravenous on Day 1 of 21 day cycles (every 3 weeks)
  Interventions: Drug: Almonertinib; Drug: Bevacizumab

INTERVENTIONS:
Drug: Almonertinib — 110 mg oral once daily
Drug: Bevacizumab — 15 mg/kg intravenous on Day 1 of 21 day cycles (every 3 weeks)

SUMMARY:
A prospective, open-label, multi-center, single-arm study of Almonertinib combined With Bevacizumab for EGFR-mutant NSCLC patients with leptomeningeal metastasis.

DETAILED DESCRIPTION:
This is a prospective, open-label, multi-center, single-arm study to evaluate the efficacy and safety of Almonertinib combined with Bevacizumab for EGFR-mutant NSCLC patients with leptomeningeal metastasis. ALL patients were treated with Almonertinib 110mg oral daily and Bevacizumab 15mg/kg intravenous every 3 weeks. Study therapy continued until disease progression, unacceptable adverse event, or withdrawal of consent.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, age in 18-75 years.
2. The Eastern Cooperative Oncology Group (ECOG) physical status score is 0-2 and has not deteriorated in the previous 2 weeks, with a minimum expected survival of 12 weeks.
3. Histologically confirmed patients with NSCLC leptomeningeal metastasis by positive cerebrospinal fluid cytological examination.
4. Tumor tissue samples or blood are confirmed to be EGFR sensitive mutations (including exon 19 deletion or L858R).
5. There must be at least one measurable extracranial lesion that has not been locally treated at the time of enrollment.
6. Females should be using adequate contraceptive measures throughout the study; should not be breastfeeding at the time of screening, during the study and until 3 months after completion of the study; and must have a negative pregnancy test prior to start of dosing if of childbearing potential or must have evidence of non-childbearing potential by fulfilling 1 of the following criteria at Screening: a) Postmenopausal defined as age more than 50 years and amenorrheic for at least 12 months following cessation of all exogenous hormonal treatments. b) Women under 50 years old would be considered postmenopausal if they have been amenorrheic for 12 months or more, following cessation of exogenous hormonal treatments, and with luteinizing hormone (LH) and follicle-stimulating hormone (FSH) levels in the postmenopausal range for the laboratory. c) Documentation of irreversible surgical sterilization by hysterectomy, bilateral oophorectomy, or bilateral salpingectomy, but not by tubal ligation.
7. Male patients should be willing to use barrier contraception (i.e., condoms).
8. For inclusion in study, patient must provide a written informed consent.

Exclusion Criteria:

1. Treatment with any of the following: a) Prior treatment with systemic anti-cancer therapy for locally advancer or metastatic NSCLC including chemotherapy, biologic therapy, immunotherapy, or any investigational drug. b) Prior treatment with an EGFR TKI. c) Major surgery (excluding placement of vascular access) within 4 weeks of the first dose of study drug. d) Radiotherapy with a limited field of radiation for palliation within 4 week of the first dose of study drug, with the exception of patients receiving radiation to > 30% of the bone marrow or with a wide field of radiation within 4 weeks of the first dose of study drug. e) Medications that are predominantly CYP3A4 strong inhibitors or inducers or sensitive substrates of CYP3A4 with a narrow therapeutic range within 7 days of the first dose of study drug.
2. Patients with other malignancies, except basal cell carcinoma and carcinoma in situ.
3. Any unresolved toxicities from prior therapy greater than Common Terminology Criteria for Adverse Events (CTCAE) Grade 1 at the time of starting study treatment, with the exception of alopecia and Grade 2, prior platinum-therapy related neuropathy.
4. Any evidence of severe or uncontrolled systemic diseases, including uncontrolled hypertension or active bleeding diatheses, which, in the Investigator's opinion, makes it undesirable for the patient to participate in the trial OR which would jeopardize compliance with the protocol such as active infection. Screening for chronic conditions is not required..
5. Refractory nausea, vomiting, or chronic gastrointestinal diseases, inability to swallow the study drug, or previous significant bowel resection that would preclude adequate absorption of Almonertinib.
6. Any of the following cardiac criteria: a) Mean resting corrected QT interval (QTc) > 470 ms obtained from 3 electrocardiograms (ECGs), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF). b) Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG (e.g., complete left bundle branch block, third-degree heart block, second-degree heart block, PR interval > 250 ms). c) Any factors that increase the risk of QTc prolongation or risk of arrhythmic events, such as heart failure, hypokalemia, congenital long QT syndrome, family history of long QT syndrome, or unexplained sudden death under 40 years of age in first degree relatives or any concomitant medication known to prolong the QT interval. d) Left ventricular ejection fraction (LVEF)< 50%.
7. Inadequate bone marrow reserve or organ function, as demonstrated by any of the following laboratory values: a) Absolute neutrophil count (ANC) <1.5×10^9 / L. b) Platelet count <100×10^9 / L. c) Hemoglobin <90 g/L (<9 g/dL). d) Alanine aminotransferase > 2.5 × upper limit of normal (ULN) if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases. e) Aspartate aminotransferase (AST) > 2.5 × ULN if no demonstrable liver metastases or > 5 × ULN in the presence of liver metastases. f) Total bilirubin (TBL) > 1.5 × ULN if no liver metastases or > 3 × ULN in the presence of documented Gilbert's Syndrome (unconjugated hyperbilirubinemia) or liver metastases. g) Creatinine > 1.5 × ULN concurrent with creatinine clearance < 50 mL/min (measured or calculated by the Cockcroft-Gault equation); confirmation of creatinine clearance is only required when creatinine is > 1.5 × ULN. h) ALB <28 g/L.
8. Past medical history of interstitial lung disease, drug-induced interstitial lung disease, radiation pneumonitis that required steroid treatment, or any evidence of clinically active interstitial lung disease.
9. Women who are breastfeeding or have a positive urine or serum pregnancy test at the Screening Visit.
10. History of hypersensitivity to any active or inactive ingredient of Almonertinib, or to drugs with a similar chemical structure or class to Almonertinib.
11. Judgment by the Investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.
12. Any severe and uncontrolled ocular disease that may, in the ophthalmologist's opinion, present a specific risk to the patient's safety.
13. Any disease or condition that, in the opinion of the Investigator, would compromise the safety of the patient or interfere with study assessments.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 69 (Estimated)
Dates: Start 2021-07 (Estimated); Primary Completion 2024-03 (Estimated); Study Completion 2025-03 (Estimated)

PRIMARY OUTCOMES:
Overall Survival (OS) | From date of enrollment until the date of death, up to 2 years
  OS is the time from the date of enrollment until death due to any cause

SECONDARY OUTCOMES:
Time to Symptom Resolution | From baseline, then every 3 weeks, up to 2 years
  Time to symptom resolution is the time from first drug dosage date (C1D1) until the date of symptom resolution
Progression Free Survival (PFS) | From baseline, then every 6 weeks, up to 2 years
  PFS is the time from date of enrollment until the date of PD (by investigator assessment) or death
Objective Response Rate (ORR) | From baseline, then every 6 weeks, up to 2 years
  ORR is the proportion of patients with a best overall response of complete response or partial response (CR+PR)
Disease Control Rate (DCR) | From baseline, then every 6 weeks, up to 2 years
  DCR is the proportion of patients with a best overall response of complete response, partial response or stable disease(CR+PR+SD)
Duration of Response (DoR) | From baseline, then every 6 weeks, up to 2 years
  DoR is the time from date of first documented response until the date of PD (by investigator assessment) or death
Intracranial Progression Free Survival (iPFS) | From baseline, then every 6 weeks, up to 2 years
  Intracranial progression-free survival
Intracranial Objective Response Rate (iORR) | From baseline, then every 6 weeks, up to 2 years
  Intracranial objective response rate
Intracranial Disease Control Rate (iDCR) | From baseline, then every 6 weeks, up to 2 years
  Intracranial disease control rate
Intracranial Duration of Response (iDoR) | From baseline, then every 6 weeks, up to 2 years
  Intracranial duration of response
Extracranial Progression Free Survival (ePFS) | From baseline, then every 6 weeks, up to 2 years
  Extracranial progression-free survival
Extracranial Objective Response Rate (eORR) | From baseline, then every 6 weeks, up to 2 years
  Extracranial objective response rate
Extracranial Disease Control Rate (eDCR) | From baseline, then every 6 weeks, up to 2 years
  Extracranial disease control rate
Extracranial Duration of Response (eDoR) | From baseline, then every 6 weeks, up to 2 years
  Extracranial duration of response
Assess the safety of Almonertinib Combined With Bevacizumab | From baseline, then every 3 weeks, up to 2 years
  Number of adverse events (AEs)/serious adverse events (SAEs)

OTHER OUTCOMES:
Evaluate the correlation between the results of CSF genetic testing and drug resistance mechanisms | CSF samples will be collected on Cycle 1 Day 1, Cycle 2 Day 1 and within one week after disease progression (each cycle is 21 days)
  Evaluate the correlation between the results of CSF genetic testing and drug resistance mechanisms

CONTACTS AND LOCATIONS:
Overall Officials: Liu Anwen, PhD, Study Director — Second Affiliated Hospital of Nanchang University
Locations (1):
- The Second Afiliated Hospital of Nanchang University, Nanchang, Jiangxi, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Pisters KM, Le Chevalier T. Adjuvant chemotherapy in completely resected non-small-cell lung cancer. J Clin Oncol. 2005 May 10;23(14):3270-8. doi: 10.1200/JCO.2005.11.478. PMID 15886314
- [Result] Bonomi PD. Implications of key trials in advanced nonsmall cell lung cancer. Cancer. 2010 Mar 1;116(5):1155-64. doi: 10.1002/cncr.24815. PMID 20087963
- [Result] Gahr S, Stoehr R, Geissinger E, Ficker JH, Brueckl WM, Gschwendtner A, Gattenloehner S, Fuchs FS, Schulz C, Rieker RJ, Hartmann A, Ruemmele P, Dietmaier W. EGFR mutational status in a large series of Caucasian European NSCLC patients: data from daily practice. Br J Cancer. 2013 Oct 1;109(7):1821-8. doi: 10.1038/bjc.2013.511. Epub 2013 Sep 3. PMID 24002608
- [Result] Maemondo M, Inoue A, Kobayashi K, Sugawara S, Oizumi S, Isobe H, Gemma A, Harada M, Yoshizawa H, Kinoshita I, Fujita Y, Okinaga S, Hirano H, Yoshimori K, Harada T, Ogura T, Ando M, Miyazawa H, Tanaka T, Saijo Y, Hagiwara K, Morita S, Nukiwa T; North-East Japan Study Group. Gefitinib or chemotherapy for non-small-cell lung cancer with mutated EGFR. N Engl J Med. 2010 Jun 24;362(25):2380-8. doi: 10.1056/NEJMoa0909530. PMID 20573926
- [Result] Burtness B, Anadkat M, Basti S, Hughes M, Lacouture ME, McClure JS, Myskowski PL, Paul J, Perlis CS, Saltz L, Spencer S. NCCN Task Force Report: Management of dermatologic and other toxicities associated with EGFR inhibition in patients with cancer. J Natl Compr Canc Netw. 2009 May;7 Suppl 1:S5-21; quiz S22-4. doi: 10.6004/jnccn.2009.0074. PMID 19470276
- [Result] Liao BC, Lee JH, Lin CC, Chen YF, Chang CH, Ho CC, Shih JY, Yu CJ, Yang JC. Epidermal Growth Factor Receptor Tyrosine Kinase Inhibitors for Non-Small-Cell Lung Cancer Patients with Leptomeningeal Carcinomatosis. J Thorac Oncol. 2015 Dec;10(12):1754-61. doi: 10.1097/JTO.0000000000000669. PMID 26334749
- [Result] Li YS, Jiang BY, Yang JJ, Tu HY, Zhou Q, Guo WB, Yan HH, Wu YL. Leptomeningeal Metastases in Patients with NSCLC with EGFR Mutations. J Thorac Oncol. 2016 Nov;11(11):1962-1969. doi: 10.1016/j.jtho.2016.06.029. Epub 2016 Aug 15. PMID 27539328
- [Result] Wu YL, Ahn MJ, Garassino MC, Han JY, Katakami N, Kim HR, Hodge R, Kaur P, Brown AP, Ghiorghiu D, Papadimitrakopoulou VA, Mok TSK. CNS Efficacy of Osimertinib in Patients With T790M-Positive Advanced Non-Small-Cell Lung Cancer: Data From a Randomized Phase III Trial (AURA3). J Clin Oncol. 2018 Sep 10;36(26):2702-2709. doi: 10.1200/JCO.2018.77.9363. Epub 2018 Jul 30. PMID 30059262
- [Result] Yang JCH, Kim SW, Kim DW, Lee JS, Cho BC, Ahn JS, Lee DH, Kim TM, Goldman JW, Natale RB, Brown AP, Collins B, Chmielecki J, Vishwanathan K, Mendoza-Naranjo A, Ahn MJ. Osimertinib in Patients With Epidermal Growth Factor Receptor Mutation-Positive Non-Small-Cell Lung Cancer and Leptomeningeal Metastases: The BLOOM Study. J Clin Oncol. 2020 Feb 20;38(6):538-547. doi: 10.1200/JCO.19.00457. Epub 2019 Dec 6. PMID 31809241
- [Result] Saboundji K, Auliac JB, Perol M, Francois G, Janicot H, Marcq M, Dubos-Arvis C, Renault A, Guisier F, Odier L, Gervais R, Chouaid C. Efficacy of Osimertinib in EGFR-Mutated Non-Small Cell Lung Cancer with Leptomeningeal Metastases Pretreated with EGFR-Tyrosine Kinase Inhibitors. Target Oncol. 2018 Aug;13(4):501-507. doi: 10.1007/s11523-018-0581-2. PMID 30039345
- [Result] Nanjo S, Hata A, Okuda C, Kaji R, Okada H, Tamura D, Irie K, Okada H, Fukushima S, Katakami N. Standard-dose osimertinib for refractory leptomeningeal metastases in T790M-positive EGFR-mutant non-small cell lung cancer. Br J Cancer. 2018 Jan;118(1):32-37. doi: 10.1038/bjc.2017.394. Epub 2017 Nov 30. PMID 29190637
- [Result] Hu X, Chen W, Li X, Zhao C, Zhang C, Xiong F, Wu H. Clinical efficacy analysis of Osimertinib treatment for a patient with leptomeningeal metastasis of EGFR+ non-small cell lung cancer without the T790M mutation. Ann Palliat Med. 2019 Nov;8(5):525-531. doi: 10.21037/apm.2019.10.13. PMID 31865717
- [Result] Seto T, Kato T, Nishio M, Goto K, Atagi S, Hosomi Y, Yamamoto N, Hida T, Maemondo M, Nakagawa K, Nagase S, Okamoto I, Yamanaka T, Tajima K, Harada R, Fukuoka M, Yamamoto N. Erlotinib alone or with bevacizumab as first-line therapy in patients with advanced non-squamous non-small-cell lung cancer harbouring EGFR mutations (JO25567): an open-label, randomised, multicentre, phase 2 study. Lancet Oncol. 2014 Oct;15(11):1236-44. doi: 10.1016/S1470-2045(14)70381-X. Epub 2014 Aug 27. PMID 25175099
- [Result] Saito H, Fukuhara T, Furuya N, Watanabe K, Sugawara S, Iwasawa S, Tsunezuka Y, Yamaguchi O, Okada M, Yoshimori K, Nakachi I, Gemma A, Azuma K, Kurimoto F, Tsubata Y, Fujita Y, Nagashima H, Asai G, Watanabe S, Miyazaki M, Hagiwara K, Nukiwa T, Morita S, Kobayashi K, Maemondo M. Erlotinib plus bevacizumab versus erlotinib alone in patients with EGFR-positive advanced non-squamous non-small-cell lung cancer (NEJ026): interim analysis of an open-label, randomised, multicentre, phase 3 trial. Lancet Oncol. 2019 May;20(5):625-635. doi: 10.1016/S1470-2045(19)30035-X. Epub 2019 Apr 8. PMID 30975627
- [Result] Nakagawa K, Garon EB, Seto T, Nishio M, Ponce Aix S, Paz-Ares L, Chiu CH, Park K, Novello S, Nadal E, Imamura F, Yoh K, Shih JY, Au KH, Moro-Sibilot D, Enatsu S, Zimmermann A, Frimodt-Moller B, Visseren-Grul C, Reck M; RELAY Study Investigators. Ramucirumab plus erlotinib in patients with untreated, EGFR-mutated, advanced non-small-cell lung cancer (RELAY): a randomised, double-blind, placebo-controlled, phase 3 trial. Lancet Oncol. 2019 Dec;20(12):1655-1669. doi: 10.1016/S1470-2045(19)30634-5. Epub 2019 Oct 4. PMID 31591063
- [Result] Lu ZQ, Cai J, Wang X, Wei JP, Zeng ZM, Huang L, Liu AW. Osimertinib combined with bevacizumab for leptomeningeal metastasis from EGFR-mutation non-small cell lung cancer: A phase II single-arm prospective clinical trial. Thorac Cancer. 2021 Jan;12(2):172-180. doi: 10.1111/1759-7714.13738. Epub 2020 Nov 17. PMID 33205587
- [Result] Matsumoto S, Takahashi K, Iwakawa R, Matsuno Y, Nakanishi Y, Kohno T, Shimizu E, Yokota J. Frequent EGFR mutations in brain metastases of lung adenocarcinoma. Int J Cancer. 2006 Sep 15;119(6):1491-4. doi: 10.1002/ijc.21940. PMID 16642476
- [Result] Lynch TJ, Bell DW, Sordella R, Gurubhagavatula S, Okimoto RA, Brannigan BW, Harris PL, Haserlat SM, Supko JG, Haluska FG, Louis DN, Christiani DC, Settleman J, Haber DA. Activating mutations in the epidermal growth factor receptor underlying responsiveness of non-small-cell lung cancer to gefitinib. N Engl J Med. 2004 May 20;350(21):2129-39. doi: 10.1056/NEJMoa040938. Epub 2004 Apr 29. PMID 15118073
- [Result] Paez JG, Janne PA, Lee JC, Tracy S, Greulich H, Gabriel S, Herman P, Kaye FJ, Lindeman N, Boggon TJ, Naoki K, Sasaki H, Fujii Y, Eck MJ, Sellers WR, Johnson BE, Meyerson M. EGFR mutations in lung cancer: correlation with clinical response to gefitinib therapy. Science. 2004 Jun 4;304(5676):1497-500. doi: 10.1126/science.1099314. Epub 2004 Apr 29. PMID 15118125